CLINICAL TRIAL: NCT02814032
Title: Differences Protein Expression in Papillary Thyroid Carcinoma
Brief Title: Proteomics of Papillary Thyroid Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Inner Mongolia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: AHInnerMongolia-Thyroid-02
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Papillary Thyroid Carcinoma
Keywords: proteomic; cervical lymph node metastasis
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- PTC group 1: papillary thyroid carcinoma patients with cervical lymph node metastasis
- PTC group 2: papillary thyroid carcinoma patients without cervical lymph node metastasis
- Positive control group: benign disease
- Negative control group: histologically normal

SUMMARY:
Thyroid carcinoma is the common endocrine system malignant neoplasm. At present it has become the malignant neoplasm of fastest growing incidence rate. More than 85% thyroid carcinoma is papillary thyroid carcinoma. Cervical lymph node metastasis is common in papillary thyroid carcinoma patients. This study aim to reveal protein expression differences between papillary thyroid carcinoma with cervical lymph node metastasis and without cervical lymph node metastasis.

DETAILED DESCRIPTION:
1. Object: Patients aged 18-65 years; newly diagnosed papillary thyroid carcinoma with cervical lymph node metastasis and without cervical lymph node metastasis and undergone thyroidectomy according to the China thyroid association guidelines for the Management of thyroid nodule and thyroid cancer.
2. Clinical information, examination data: Information is obtained from medical record abstraction.
3. Samples: Fresh frozen thyroid tissues from each sample group(normal histology, benign disease, papillary thyroid carcinoma with cervical lymph node metastasis, papillary thyroid carcinoma without cervical lymph node metastasis ).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed papillary thyroid carcinoma.
* Undergo thyroidectomy according to the China thyroid association guidelines forthe Management of thyroid nodule and thyroid cancer.

Exclusion Criteria:

* Current substance abuse/dependence.
* Daily tobacco and alcohol use.
* Whole neck irradiation or surgery.
* Prior cancer diagnosis or chemotherapy treatment.
* Active autoimmune disorder.
* Uncontrolled allergic condition or asthma.
* Chronic use of oral steroid medication.
* Hormone therapy (estrogen, progestin compounds).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years; newly diagnosed papillary thyroid carcinoma with cervical lymph node metastasis and without cervical lymph node metastasis and undergone thyroidectomy according to the China thyroid association guidelines for the Management of thyroid nodule and thyroid cancer.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2016-06; Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
differences in protein expression | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shan Jin, PhD, Study Director — The Affiliated Hospital of Inner Mongolia Medical University
Locations (1):
- Shan Jin, Hohhot, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gharib H, Papini E. Thyroid nodules: clinical importance, assessment, and treatment. Endocrinol Metab Clin North Am. 2007 Sep;36(3):707-35, vi. doi: 10.1016/j.ecl.2007.04.009. PMID 17673125
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Brown LM, Helmke SM, Hunsucker SW, Netea-Maier RT, Chiang SA, Heinz DE, Shroyer KR, Duncan MW, Haugen BR. Quantitative and qualitative differences in protein expression between papillary thyroid carcinoma and normal thyroid tissue. Mol Carcinog. 2006 Aug;45(8):613-26. doi: 10.1002/mc.20193. PMID 16788983
- [Background] Sofiadis A, Becker S, Hellman U, Hultin-Rosenberg L, Dinets A, Hulchiy M, Zedenius J, Wallin G, Foukakis T, Hoog A, Auer G, Lehtio J, Larsson C. Proteomic profiling of follicular and papillary thyroid tumors. Eur J Endocrinol. 2012 Apr;166(4):657-67. doi: 10.1530/EJE-11-0856. Epub 2012 Jan 24. PMID 22275472